CLINICAL TRIAL: NCT02186405
Title: Effects of Levothyroxine Treatment on Hemodynamic and Isotopic Renal Functions in Subclinical Hypothyroidism
Brief Title: Effects of Levothyroxine Treatment on Hemodynamic and Renal Functions in Subclinical Hypothyroidism
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No patient corresponding to inclusion criteria couldn't be enrolled in the study
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-AOI-03
Record Dates: First submitted 2014-07-08; First posted 2014-07-10 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Subclinical hypothyroïdism
MeSH Terms: interventions — Thyroxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LEVOTHYROXINE (Experimental): administration of levothyroxine
  Interventions: Drug: LEVOTHYROXINE

INTERVENTIONS:
Drug: LEVOTHYROXINE — administration of levothyroxine

SUMMARY:
Renal and cardiovascular effects of subclinical hypothyroidism, defined by a high TSH and normal T4 are less known and the indications for treatment of subclinical hypothyroidism are subject to controversies.

The investigators propose to assess whether the hormone replacement for subclinical hypothyroidism in patients with chronic kidney disease is beneficial for hemodynamic and renal functions and which mechanisms are involved.

Isotopic measurements of glomerular filtration and renal blood flow and an hemodynamic evaluation by transthoracic echocardiography and flow-mediated vasodilation will be carried out before and 6 months after substitution.

DETAILED DESCRIPTION:
Animal experimental hypothyroidism is associated with renal and hemodynamic abnormalities. In human, exact measurements of GFR showed a decline in GFR after thyroidectomy and an increase in GFR and renal blood flow after hormone replacement. Renal and cardiovascular effects of subclinical hypothyroidism, defined by a high TSH and normal T4 are less known and the indications for treatment of subclinical hypothyroidism are subject to controversies. A retrospective study suggests that treatment of subclinical hypothyroidism may slow the degradation rate of renal function estimated by MDRD. However, the potential hemodynamic benefit of treatment has not yet been studied.

The investigators propose to assess whether the hormone replacement for subclinical hypothyroidism in patients with chronic kidney disease is beneficial for hemodynamic and renal functions and which mechanisms are involved.

Isotopic measurements of glomerular filtration and renal blood flow and an hemodynamic evaluation by transthoracic echocardiography and flow-mediated vasodilation will be carried out before and 6 months after substitution. This open prospective study will include 16 patients in order to detect an increase of 1.2 standard deviation for the measured glomerular filtration.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years
* chronic kidney disease
* subclinical hypothyroidism

non-inclusion Criteria:

* insulin-dependent diabetes
* dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2016-10 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
KIDNEY CLEARANCE | Before treatment and 6 months after treatment
  (51)Cr-EDTA clearance after 6 months of hormonal replacement

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume FAVRE, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- Nephrology Department, Nice, France